CLINICAL TRIAL: NCT03533920
Title: A Single-arm, Multicenter, Open, Pivotal Clinical Trial to Evaluate the Efficacy and Safety of UNI-DEB for Unresectable Hepatocellular Carcinoma
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of UNI-DEB for Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNI-DEB-Pivotal
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Hepatocellular Carcinoma Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UNI-DEB (Experimental)
  Interventions: Device: UNI-DEB

INTERVENTIONS:
Device: UNI-DEB — Applicate the TACE with UNI-DEB to unresectable hepatocellular carcinoma patient

SUMMARY:
Pivotal Clinical Trial to Evaluate the Efficacy and Safety of UNI-DEB for Unresectable Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years
* Diagnosis of HCC
* Unresectable asymtomatic uninodular or multinodular tumor.
* Subject who maintain clinically normal hepatopetal flow without main portal vein closure
* At least one measurable target lesion by CT or MRI which 10 mm or more and 100 mm or less.
* ECOG Performance Status of 0 or 1.
* Child-Pugh class A or B
* Life expectancy of at least 6 months.

Exclusion Criteria:

* Another primary tumour, with the exception of conventional basal cell carcinoma or superficial bladder neoplasia
* Hepatic resection, liver transplantation or Percutaneous local treatment
* Previously received HCC related medical procedure
* Previously treated with anthracyclines
* Only measurable disease is within an area of the liver previously subjected to radiotherapy.
* Child Pugh C
* Active gastrointestinal bleeding within 6 months from screening.
* Total bilirubin > 3mg/dL
* WBC < 3,000cells/mm3
* Platelet < 50,000mm3
* Serum creatinine > 2mg/dL
* INR> 1.4
* ALT and AST > 5 times UNL
* Diffuse HCC defined as >50% tumour involvement of the whole liver.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate by independent evaluator | 4 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (8):
- South Korea (8):
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - The Catholic University of Korea, Uijeongbu ST. Mary's Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Pusan National University Hospital, Pusan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No